CLINICAL TRIAL: NCT01184924
Title: Evaluation of the Arthritis Foundation Tai Chi Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Leigh F Callahan, PhD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-1048
Record Dates: First submitted 2010-08-13; First posted 2010-08-19 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Arthritis
Keywords: Arthritis; Tai Chi
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual Care only. Usual care is defined as the care these subjects would like to seek from any health care practitioner or other program they may seek for healthy living. The subjects in this arm will be offered the AF Tai Chi intervention after an 8 week followup data collection
- Tai Chi (Experimental): Usual care plus Tai Chi. These subjects will be allowed to seek care from any health practitioner or any other programs and will receive the AF Tai Chi program for 8 weeks.
  Interventions: Behavioral: Evaluation of the Arthritis Foundation Tai Chi Program

INTERVENTIONS:
Behavioral: Evaluation of the Arthritis Foundation Tai Chi Program — The primary goal of this study is to assess the effectiveness and feasibility of the arthritis foundation (AF) Tai Chi Program for People with Arthritis. Arthritis, the most prevalent chronic condition in the US and a leading cause of disability, is characterized by chronic pain and progressive impairment of joints and soft tissues. Promoting physical activity is a key public health strategy to addressing arthritis management, but more scientific data regarding effectiveness and feasibility are need to support the promotion of the AF Tai Chi Program as an exercise intervention for people with arthritis. Participants will be randomly assigned to the intervention or delayed control arm of the study.
  Arms: Tai Chi

SUMMARY:
The primary goal of this study is to assess the effectiveness and feasibility of the arthritis foundation (AF) Tai Chi Program for People with Arthritis. Arthritis, the most prevalent chronic condition in the US and a leading cause of disability, is characterized by chronic pain and progressive impairment of joints and soft tissues. Promoting physical activity is a key public health strategy to addressing arthritis management, but more scientific data regarding effectiveness and feasibility are need to support the promotion of the AF Tai Chi Program as an exercise intervention for people with arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Self-Reported doctor diagnosed arthritis
* Age 18 years or older
* Able to move independently without assistance

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Cognitive impairment
* Serious medical conditions: History of MI, stroke, prescribed beta-blockers, surgery in past 6 months, uncontrolled hypertension, chest pain, diabetes mellitus
* Severe impairment of physical functioning
* Participation in Tai Chi exercise in last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Arthritis symptoms. | Baseline , 8 weeks from baseline assessment, 1 year from baseline asssessment
  Arthritis symptoms include pain, stiffness and fatigue as measured using a 10 cm Visual Analog Scale (VAS)
Health Assessment Questionnaire (HAQ) | Baseline, 8 weeks from baseline assessment, 1 year from baseline asssessment
  The disability scale of the HAQ will be used to assess physical functioning and disease progression. As a disease specific measure it is used in much of the rheumatological literature. It includes items querying 20 specific activities of daily living in 8 domains (dressing, arising, eating, walking, hygiene, activities, ready, grip) and adjusts scores based on the use of assistive devices. The HAQ is scored from 0 to 3, with 0 representing no disability and 3 representing maximum disability.
Arthritis Self Efficacy (ASE) | Baseline, 8 weeks from baseline assessment, 1 year from baseline asssessment
  Self-efficacy for managing arthritis will be assessed using two subscales from the Arthritis Self Efficacy Scale developed by Lorig and colleagues. The scale assess the degree to which an individual feels confident about his or her ability to manage his or her arthritis including decreasing pain, keeping pain from interfering with normal activities, and dealing with frustration of having arthritis. The pain subscale (5 items) and the other symptoms subscale (6 items) will be used. The items are scored on a Likert-type scale with 0= "very uncertain" and 100= "very certain"
Falls Surveillance | Baseline, 8 weeks from baseline assessment, 16 weeks from baseline assessment.
  Adapting a previously used method to the particular schedule of this protocol, both intervention and control participants will be given a "falls calendar" at baseline and instructed to record each day for 16 weeks if they had a fall. Falls are defined as "unintentially coming to rest on the floor or ground". This record will cover the intervention group through the 8 week Tai Chi course and or an 8 week follow up period. The control group record will cover the 8 weeks before Tai Chi and during the delayed Tai Chi course. The calendars will be mailed in after completion.
50 Foot Walk Test | Baseline, 8 weeks from baseline assessment
  This is an objective measure of submaximal walking function in older adults with arthritis. It was developed to be an outcome measure of physical function for subjects participating in pharmacological clinical trials of arthritis medications.
Multidirectional Reach Test | Baseline, 8 weeks from baseline assessment
  This test is a balance test developed to study falls in the elderly. Performed while either sitting or standing, (feet comfortably apart) subjects reach in either a forward, backward or sideways direction. Distances reached are measured in inches. The tool has high inter-rater reliability (ICC=.99) and test-retest reliability (ICC-.98) The tool has been shown to have a concurrent validity with the Berg Balance and Timed up and Go Tests.
Timed Chair Stands Test | Baseline, 8 weeks from baseline assessment
  This test is a functional strength test. It tests the coordinated control of the body's center of mass in order to maintain dynamic balance as the base of support is transitioned from sitting on a chair with feet on the ground (3-point) to standing (2 point). Test-retest reliability has been show to be ICC=.84 for men and .92 for women. It has also shown to have concurrent validity with maximum weight adjusted leg press performance.
Single Leg Stance (SLS) | Baseline, 8 weeks from baseline assessment
  This is a timed test which has been correlated with amplitude and speed of sway in individuals without disease. The ability to maintain SLS generally decreases with increasing age. The test is performed with eyes open, and subjects stand on one leg while placing arms across their chest.

SECONDARY OUTCOMES:
Secondary outcomes are psychosocial measures. | Baseline, 8 weeks from baseline assessment, 1 year from baseline assessment
  Psychosocial measures include: Rheumatology Attitudes Index (RAI, helplessness)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh F Callahan, PhD, Principal Investigator — University of North Carolina at Chapel Hill, Thurston Arthritis Research Center